CLINICAL TRIAL: NCT01495429
Title: A Phase III Study of Peripherally Inserted Versus Centrally Inserted Central Venous Catheters in the Neurological Intensive Care Unit
Brief Title: Peripherally Inserted Versus Centrally Inserted Central Venous Catheters in the Neurological Intensive Care
Acronym: PICNIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey J Fletcher, Study PI, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00050032
Record Dates: First submitted 2011-12-13; First posted 2011-12-20 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Venous Thrombosis
Keywords: catheter related large vein thrombosis; upper extremity deep venous thrombosis; central venous catheters; upper extremity catheter related large vein thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Central Venous Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PICC line (Peripherally) (Experimental): placement of a picc line
  Interventions: Procedure: Central venous catheter
- CICVC (central insertion) (Active Comparator): placement of a centrally inserted central venous catheter
  Interventions: Procedure: Central venous catheter

INTERVENTIONS:
Procedure: Central venous catheter — Placement of a peripherally inserted central venous catheter
  Arms: PICC line (Peripherally)
Procedure: Central venous catheter — Placement of a centrally inserted central venous catheter
  Arms: CICVC (central insertion)

SUMMARY:
The investigators aim to compare the complications between centrally and peripherally inserted central venous catheters in neurological intensive care unit patients. The study hypothesis is that peripherally inserted catheters will have more cumulative complications due to venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* all patients age > 18, admitted to the neurological ICU who are require a de novo central venous catheter as standard of care and in which a double lumen 5f PICC or CICVC (triple lumen, 7f) are acceptable for the indication.
* the patients must be expected to survive and need a central venous catheter for at least 7 days.

Exclusion Criteria:

* prisoner
* age < 18
* expected to die or have care withdrawn prior to ICU day 7
* requiring an emergent central venous catheter
* suspected bacteremia
* recent central venous catheter within the last 30 days
* patients who are not a candidate for bedside placement of either a CICVC or PICC line
* patients with renal insufficiency with creatinine level greater than 3.0 mg/dL (265.2 m mol/L) or who were undergoing hemodialysis
* patients requiring a central venous catheter for prolonged antibiotic therapy\
* patient who the treating clinician feels clearly needs one particular type of catheter over the other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The composite of death or catheter related large vein thrombosis | 15 days

SECONDARY OUTCOMES:
Cumulative catheter related complications until discharge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Fletcher, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan